CLINICAL TRIAL: NCT05334368
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of Depemokimab in Adults With Hypereosinophilic Syndrome (HES)
Brief Title: Depemokimab in Participants With Hypereosinophilic Syndrome, Efficacy, and Safety Trial
Acronym: DESTINY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 217013
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Hypereosinophilic Syndrome
Keywords: Depemokimab; Hypereosinophilic Syndrome; DESTINY; Monoclonal antibody; Anti-interleukin -5
MeSH Terms: conditions — Hypereosinophilic Syndrome

STUDY DESIGN:
Intervention Model Description: This is a randomized, placebo-controlled, double-blind, parallel group, multicenter study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a double-blind study with respect to allocation of depemokimab or placebo to participants. All site staff, participants, and investigator will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Depemokimab (Experimental): All participants in this arm will receive depemokimab.
  Interventions: Drug: Depemokimab
- Placebo (Placebo Comparator): All participants in this arm will receive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Depemokimab — Depemokimab will be administered.
  Arms: Depemokimab
Other: Placebo — Matching placebo will be administered.
  Arms: Placebo

SUMMARY:
This is a 52-week, randomized, placebo-controlled, double-blind, parallel group, multicenter study of depemokimab in adults with uncontrolled HES receiving standard of care (SoC) therapy.

The study will recruit patients with a confirmed diagnosis of HES and who are on stable HES therapy for at least 4 weeks prior to randomization (Visit 2). Eligible participants must have uncontrolled HES with a history of repeated flare (≥2 flares in the previous 12 months) and blood eosinophil count of ≥1,000 cells/ microliter (μL) during Screening. Historical HES flares are defined as documented HES-related worsening of clinical symptoms or blood eosinophil counts requiring an escalation in therapy.

Participants who meet the inclusion and exclusion criteria will be randomized in a 2:1 ratio to receive either depemokimab or placebo while continuing their SoC HES therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are greater than or equal (>=) 40 kilogram (kg) at Screening Visit 1.
* Participants who have a documented diagnosis of HES prior to Visit 2.
* A history of 2 or more HES flares within the past 12 months prior to Visit 1.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies: a) woman of non-childbearing potential (WONCBP) Or b) woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective, with a failure rate of less than (<) 1 percentage (%).
* Capable of giving signed informed consent.

Exclusion Criteria:

* Participants with HES disease manifestations which in the opinion of the investigator may put the participant at unacceptable risk from study participation or confound interpretation of efficacy or safety data.
* Participants with chronic or ongoing active infections requiring systemic treatment or a pre-existing parasitic infestation within 6 months prior to Visit 1.
* Participants with a known immunodeficiency (e.g., Human Immunodeficiency Virus [HIV]), other than that explained by the use of OCS or other therapy taken for HES.
* Participants with a history of or current lymphoma.
* Participants with current malignancy or previous history of cancer in remission for less than 5 years prior to Visit 1. Participants that had localized carcinoma (i.e., basal or squamous cell) of the skin which was resected for cure will not be excluded.
* Participants with a haematologic malignancy with hypereosinophilia in which HES is not the primary diagnosis, e.g., chronic myeloid leukaemia, myelodysplastic syndrome, chronic eosinophilic leukaemia-not otherwise specified.
* Cirrhosis or current unstable liver or biliary disease per investigator assessment.
* Participants who have severe or clinically significant cardiovascular disease uncontrolled with standard treatment.
* Participants with current diagnosis of vasculitis.
* Hypereosinophila with no clinical symptoms and/or proof of organ dysfunction.
* Clinical diagnosis of Eosinophilic granulomatosis with polyangiitis (EGPA).
* Participants with an allergy/ intolerance to a monoclonal antibody or biologic, or any of the excipients of the investigational product.
* Participants who have a previous documented failure with anti-interleukin (IL)-5/5R therapy.
* Participants who have received monoclonal antibodies (mAb) within 30 days or 5 half-lives, whichever is longer, prior to Visit 1.
* Participants who test positive for the FIP1L1-PDGFRα fusion gene.
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) ≥450 milliseconds (msec) or QTcF ≥480 msec for participants with Bundle Branch Block at Screening Visit 1.
* Participants who are not responsive to OCS based on clinical response or blood eosinophil counts in the opinion of the Investigator.
* Participants who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2028-12-19 (Estimated); Study Completion 2028-12-19 (Estimated)

PRIMARY OUTCOMES:
Frequency of HES flares | Up to 52 weeks
  A HES flare is defined as either: a HES-related clinical manifestation based on a physician documented change in clinical signs or symptoms resulting in the need for the following : An increase in the maintenance systemic corticosteroid dose by at least 10 mg/day (prednisone/prednisolone equivalent) for at least 5 days, and/or an increase in or addition of any cytotoxic and/or immunosuppressive HES therapy.
  OR 2 or more courses of blinded active oral corticosteroid (OCS) during the intervention period. The frequency of HES flares will be calculated for each participant as the number of unique starting dates for HES flares.

SECONDARY OUTCOMES:
Time to first HES flare | Up to 52 weeks
  The time to first HES flare will be calculated from the date of first dose of study intervention and the start date of the HES flare. Time to the first HES flare will be assessed and reported in days.
Number of participants with at least one HES flare during the 52-week study intervention period | Up to 52 weeks
Change from Baseline to Week 52 in weekly average score of Brief Fatigue Inventory (BFI) item 3 (worst fatigue in last 24 hours) | Baseline and up to Week 52
  The BFI is a tool developed for the rapid assessment of fatigue severity for use in both clinical Screening and clinical trials. The BFI has 9 items. The participant should rate their average and worst fatigue levels over the previous 24 hours using a numeric rating scale anchored with 0 (no fatigue/interference) and 10 (as bad as you can imagine/completely interferes) numeric rating scales

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (82):
- United States (11):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Southfield, Michigan
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Salt Lake City, Utah
- Argentina (5):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Florida
  - GSK Investigational Site, La Plata
  - GSK Investigational Site, Mar del Plata
  - GSK Investigational Site, Quilmes
- GSK Investigational Site, Garran, Australian Capital Territory, Australia
- GSK Investigational Site, Brussels, Belgium
- Brazil (4):
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Blumenau
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, Sorocaba
- Canada (2):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
- China (8):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Harbin
  - GSK Investigational Site, Nanchang
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Suzhou
  - GSK Investigational Site, Wuhan
- Czechia (4):
  - GSK Investigational Site, Brno-Bohunice
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Ústí nad Labem
- GSK Investigational Site, Odense C, Denmark
- Germany (2):
  - GSK Investigational Site, Bad Bramstedt
  - GSK Investigational Site, Mannheim
- Greece (2):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Rio Patras
- GSK Investigational Site, Pokfulam, Hong Kong
- Israel (2):
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Tel Aviv
- Italy (9):
  - GSK Investigational Site, Bologna
  - GSK Investigational Site, Catania
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Novara
  - GSK Investigational Site, Pavia
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Treviso
  - GSK Investigational Site, Verona
- Japan (9):
  - GSK Investigational Site, Aomori
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Wakayama
  - GSK Investigational Site, Yamanashi
- Mexico (3):
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Monterrey
  - GSK Investigational Site, Veracruz
- Poland (2):
  - GSK Investigational Site, Chęciny
  - GSK Investigational Site, Lodz
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
- South Korea (5):
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Kangwondo
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon Kyunggi-do
- Spain (7):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pozuelo de AlarcOn Madr
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Zaragoza
- GSK Investigational Site, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- See also: Related Info — https://gskdestinystudy.com/?utm_source=ctgov